CLINICAL TRIAL: NCT01140607
Title: Phase I Safety and Pharmacokinetic Study of XRP6258 (Cabazitaxel) In Advanced Solid Tumor Patients With Varying Degrees of Hepatic Impairment
Brief Title: Safety and Pharmacokinetic Study of Cabazitaxel in Patients With Advanced Solid Tumors and Liver Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POP6792; U1111-1116-5845 (Other: UTN)
Record Dates: First submitted 2010-05-28; First posted 2010-06-09 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — cabazitaxel; XRP6258

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Cohort 1: normal hepatic function: cabazitaxel (Experimental): cabazitaxel 25mg/m^2
  IV infusion of Cabazitaxel is given over 1 hour on Day 1 of each cycle (every 3 weeks).
  Interventions: Drug: Cabazitaxel (XRP6258)
- Cohort 2: mild hepatic impairment : cabazitaxel (Experimental): cabazitaxel 20mg/m^2
  IV infusion of Cabazitaxel is given over 1 hour on Day 1 of each cycle (every 3 weeks).
  Interventions: Drug: Cabazitaxel (XRP6258)
- Cohort 3: moderate hepatic impairment: cabazitaxel (Experimental): cabazitaxel 10mg/m^2
  IV infusion of Cabazitaxel is given over 1 hour on Day 1 of each cycle (every 3 weeks).
  Interventions: Drug: Cabazitaxel (XRP6258)
- Cohort 4: severe hepatic impairment: cabazitaxel (Experimental): cabazitaxel 5 mg/m^2 or 10mg/m^2
  IV infusion of Cabazitaxel is given over 1 hour on Day 1 of each cycle (every 3 weeks).
  Interventions: Drug: Cabazitaxel (XRP6258)
- Cohort 5: normal hepatic function: cabazitaxel and midazolam (Experimental): cabazitaxel 25mg/m^2
  IV infusion of Cabazitaxel is given over 1 hour on Day 1 of each cycle (every 3 weeks).
  Midazolam is given orally in single dosing on day -1 and day 1 (crossover)
  Interventions: Drug: Cabazitaxel (XRP6258)

INTERVENTIONS:
Drug: Cabazitaxel (XRP6258) — Pharmaceutical form:solution for infusion
  Route of administration: intravenous

SUMMARY:
Primary Objectives:

* To determine the maximum tolerated dose (MTD) and safety of Cabazitaxel when administered to advanced solid tumor patients with varying degrees of hepatic impairment
* To determine the pharmacokinetics (PKs) of Cabazitaxel in patients with varying degrees of hepatic impairment
* To correlate PK variables with pharmacodynamic (PD) safety parameters in order to guide prescribers with regard to dosing in this patient population
* To assess the effect of cabazitaxel at recommended dose of 25mg/m^2 on CYP3A enzyme activity using midazolam as probe in an additional cohort of cancer patients with normal hepatic function.

DETAILED DESCRIPTION:
The study consists of:

* a screening phase (maximum length of 21-day).
* a treatment phase with 21-day study treatment cycles. Cycle lengths may be extended up to maximum of 12 additional days in case of unresolved toxicity.

Patients continue to receive treatment until they experience, unacceptable toxicities/AEs, disease progression ,withdraw their consent, or the investigator decides to discontinue the patient, or study cut-off, whichever comes first.

* a 30-day follow-up visit after the last dose of study medication.

The cut off date is when the last patient treated has completed cycle 1 and the subsequent 30 days follow-up.

Patients may continue to be treated as long as they are benefiting from study treatment and have not met study withdrawal criteria.

ELIGIBILITY:
Inclusion criteria:

* Patients with a diagnosis of advanced, measurable or non-measurable, non-hematological cancer who have varying degrees of hepatic impairment. The cancer must be one that is either refractory to standard therapy or for which no standard therapy exists.

Exclusion criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) >2
* Life expectancy <3 months
* Need for a major surgical procedure or radiation therapy during the study
* Evidence of another active malignancy
* Prior chemotherapy, other investigational drug, biological therapy, targeted non-cytotoxic therapy and radiotherapy within 3 weeks prior to registration
* Patients with known history of Gilbert's syndrome
* Prior treatment with Cabazitaxel and a history of severe (Grade ≥3) hypersensitivity to taxanes, polysorbate-80, or to compounds with similar chemical structures
* Prior history of bone marrow transplant
* Any treatment known to induce CYP isoenzymes or to inhibit CYP3A4 activities within 2 weeks before or during the test period of the pharmacokinetic sampling. Moderate inhibitors within one week prior and during the pharmacokinetic sampling.
* Any contra-indications to midazolam, according to the applicable labeling.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2010-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLT) | cycle 1 (3 weeks)
  A clinical adverse event or a laboratory abnormality is defined as DLT when it is drug-related as assessed by the investigator and agreed upon by the study committee.

SECONDARY OUTCOMES:
Safety investigations (physical examination, vital signs and laboratory tests) | up to 30 days after the last dosing
  Physical examination includes Eastern Cooperative Oncology Group (ECOG) performance status and signs and symptoms.
  Vital signs includes weight, temperature, blood pressure and heart rate.
  Laboratory tests includes hematology, coagulation, biochemistry and urinalysis. Laboratory abnormalities are graded according to the NCI CTCAE v.4.0
Pharmacokinetic profile of Cabazitaxel (AUC, Cmax, t1/2, CL, and Vss) from plasma concentration | cycle 1 (3 weeks)
Cabazitaxel effect on CYP3A enzyme activity | single dosing on day -1 and day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (14):
- United States (14):
  - Investigational Site Number 840014, La Jolla, California
  - Investigational Site Number 840013, Loma Linda, California
  - Investigational Site Number 840020, Washington D.C., District of Columbia
  - Investigational Site Number 840016, Jacksonville, Florida
  - Investigational Site Number 840002, Tampa, Florida
  - Investigational Site Number 840017, Decatur, Illinois
  - Investigational Site Number 840003, Metairie, Louisiana
  - Investigational Site Number 840019, Baltimore, Maryland
  - Investigational Site Number 840012, Boston, Massachusetts
  - Investigational Site Number 840001, St Louis, Missouri
  - Investigational Site Number 840021, Canton, Ohio
  - Investigational Site Number 840007, Cincinnati, Ohio
  - Investigational Site Number 840010, Bethlehem, Pennsylvania
  - Investigational Site Number 840006, San Antonio, Texas